CLINICAL TRIAL: NCT04907071
Title: Intravascular Ultrasound for the Evaluation of Malperfusion Syndrome in the Setting of Acute Aortic Dissection: A Pilot Study.
Brief Title: Intravascular Ultrasound for the Evaluation of Malperfusion Syndrome in the Setting of Acute Aortic Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Karama Bayamin, Cardiac Surgery Resident, London Health Sciences Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAD IVUS
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Aortic Dissection; Perfusion; Complications
Keywords: Malperfusion; Syndrome
MeSH Terms: conditions — Aortic Dissection; Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Malperfusion Primary Cohort (Experimental): Patients presenting to hospital with AAD meeting criteria for malperfusion syndrome preoperatively which includes both components:
  * Imaging findings indicating reduced flow to the Celiac Trunk, Superior mesenteric artery, either renal artery or either iliac artery
  * Clinical stigmata of end organ ischemia (abdominal pain, distended abdomen, oliguria/anuria, reduced pulses, signs of limb ischemia) OR Laboratory findings suggestive of end organ ischemia (lactic acidosis, elevated LFTs, Elevated Creatinine, Rhabdomyolysis, Electrolyte abnormalities)
  Interventions: Device: Intravascular ultrasound 0.035 PV IVUS catheter (Volcano Therapeutics, Rancho Cordova, CA)
- Malperfusion Secondary Cohort: (Experimental): Patients who develop new clinical signs or laboratory results indicating distal malperfusion after proximal repair of the AAD is complete and proximal blood flow is redirected into the true lumen.
  * New Clinical signs include: Loss of femoral pulses, distended abdomen, reduced urine output, dusky extremities
  * New Laboratory signs include: Rising lactate (>50% above baseline), Rising Creatinine, Metabolic Acidosis, Rising LFTs
  Interventions: Device: Intravascular ultrasound 0.035 PV IVUS catheter (Volcano Therapeutics, Rancho Cordova, CA)
- No Malperfusion Cohort (Experimental): Patients presenting with AAD with no evidence of malperfusion syndrome preoperatively and postoperatively.
  Interventions: Device: Intravascular ultrasound 0.035 PV IVUS catheter (Volcano Therapeutics, Rancho Cordova, CA)

INTERVENTIONS:
Device: Intravascular ultrasound 0.035 PV IVUS catheter (Volcano Therapeutics, Rancho Cordova, CA) — The investigational 0.035 PV IVUS catheter (Volcano Therapeutics, Rancho Cordova, CA) is an over the wire catheter-based ultrasound with an 8.2-French profile at the transducer end and 7.0-French shaft diameter. This is run through a 9-French place under surface ultrasound guidance in the common femoral artery. The working length of this catheter is 90 cm, with the ability to imaging a diameter up to 60 mm.7

SUMMARY:
Aortic dissection is a life-threatening condition caused by a tear in the internal layer of major artery wall (aorta) that carries blood to all body organs, resulting in separation of the aortic wall layers (dissection). The dissected aorta compromises blood flow to any organ, and eventually leads to organ damage (Malperfusion Syndrome).

Our goal in this project is to use Intravascular Ultrasound (IVUS) to have real time assessment and confirm any evidence of malperfusion syndrome in the setting of aortic dissection after repairing the original aortic tear. IVUS is a small ultrasound (sound waves) wand that is attached to the top of a thin tube. This tube is inserted into the aorta from the groin. This device takes pictures of the aorta and its major branches, to identify problems with blood flow. Having this real-time and dynamic assessment will help to identify any malperfused organs before leaving the operating room and allow us to address the malperfusion syndrome as quickly as possible to limit complications. Without this technique, identifying the problem can take several days after surgery at which point there can be irreversible complications.

DETAILED DESCRIPTION:
Acute Type A Aortic Dissection

A Debakey acute type A aortic dissection (ATAAD) represents a lethal condition with a risk of mortality of 1% per hour and up to nearly 50% in first 48 hours if left untreated.1, 2 Traditional surgical teaching has always involved emergent repair of the proximal aortic with resection and replacement of the intima entry tear and aneurysmal tissue within the ascending aorta. This approach addresses obviates the risk of aortic rupture, proximal extension into the coronary arteries, cardiac tamponade and aortic valve insufficiency, all of which lead to mortality. However, as expertise in the field progress evidence is emerging that dealing with only the proximal extent of the dissection may still leave a significant portion of patients at risk for complications from an inability to identify and treat end-organ malperfusion.3 At Western University and London Health Sciences center our mortality rate for patients presenting the ATAAD has been reporter at 20.0%4, and is similar to that reported by the International Registry of Acute aortic Dissection (IRAD) database, with mortality rates between 16.2 and 27.4%.5,6

Malperfusion Syndrome and Aortic Rupture In the 2018 Circulation paper published by Yang et al. the University of Michigan group outline the treatment strategy for ATAAD.

In this study, all patients with an ATAAD presenting with malperfusion, but without signs of aortic rupture or cardiac tamponade, were treated first with endovascular revascularization followed by delayed open aortic repair.3 The authors report that in the second decade of their experience with this treatment model, the overall mortality dropped to 10.7%.3 When compared to our local data and that published by the IRAD group, it would appear that there are significant improvements that can be made for the treatment of these individuals. The authors report that roughly 1/3 of all patients presented with some form of malperfusion syndrome and that in this group, 87% of the deaths were attributed to organ failure from malperfusion even after fenestration and stenting. Conversely there was only a 4% risk of aortic rupture following fenestration and stenting prior to open surgical repair in this group.3 This would indicate that malperfusion is a significant cause of morbidity and mortality in these patients maybe even more so than the risk of aortic rupture in selective patients but in order to improve our outcomes, we need a better way to assess static and dynamic changes that cause malperfusion as early as possible.

Static and Dynamic Arterial Malperfusion

The concept of static and dynamic obstructions in regards to aortic blood flow, indicates the phenomenon where disruption of laminar flow due to interruption of the intimal layer in and aortic dissection, results in gradients between the true and false lumen which can shear a dissection flap over a branching vessel causing collapse of the true lumen (dynamic), or the development of thrombus within the false lumen resulting in obstruction of a branch vessel (static). Most emergent AAD repairs will involve a baseline CT scan of the chest, abdomen and pelvis, which may identify malperfusion of distal arteries shown by a lack of contrast opacification. However, this is done prior to surgical repair and not an accurate representation of perfusion after proximal surgical repair is completed. Frist of all, at the time of the initial CT scan the intimal tear is still present and flow may not be directed into the true lumen, patients blood pressures may not be controlled which can cause dynamic shifts in the intimal flap favouring either true or false lumen flow, and lastly multiple distal re-entry tears can form throughout the remaining aorta after surgical repair which also have the capability of altering arterial flow. Transesophageal echocardiogram is usually present at the time of open surgical repair, but it is limited to the ascending, arch and descending thoracic aorta and provides little information regarding flow to the visceral segments, kidneys and legs.

Intravascular Ultrasound (IVUS)

Intravascular Ultrasound (IVUS) has been used over the past several decades for the real-time assessment of vascular anatomy in a variety of clinical settings.7 Standard IVUS catheters typically use a 9-French delivery sheath and are run over a 0.035-inch guidewire. The device transducer emits and receives signals at varying frequencies to produce a 360̊ axial image. As surgeons are becoming more familiar with this technology and developing the skill set necessary to use the equipment, including the real-time acquisition and interpretation of images, it permits the full evaluation of the thoracoabdominal aorta including size, tortuosity, and calcification. In the setting of an AAD, IVUS can provide real-time data under physiologic conditions following open proximal repair to indicate the presence of distal re-entry tears, compression of the true lumen and malperfusion to aortic branches. It also, can be used intraoperatively to confirm resolution of malperfusion to the visceral segments and legs after proximal flow is reinsituted into the true lumen.

Study Rationale

As noted above, AAD is a lethal condition that every cardiovascular surgeon is faced with at some point in their career. Although the outcomes at LHSC have been historically very good and are on par with or better than the existing IRAD data, looking at other institutions who have more advanced approaches, there appears to be some room to improve our outcomes even further. We believe that emergent repair of the proximal extent of the AAD, which is the current standard at LHSC, results in stabilization of the aortic valve, protects coronary flow, relieves cardiac tamponade and reduces the risk of aortic rupture. However, this approach leaves patients at risk for distal malperfusion due to distal re-entry tears, patent false lumens and thrombus formation, creating both dynamic and static obstruction. Intraoperative IVUS evaluation would therefore allow for the assessment of distal perfusion immediately following proximal repair in order to identify malperfusion and adjust treatment accordingly to prevent damage from prolonged end-organ ischemia. The purpose of this study is to test the safety and efficacy of intraoperative IVUS immediately following open surgical repair.

Device Description

The study devices are intended to improve outcomes for patients presenting with malperfusion syndrome in the setting of ATAAD. Every subject in the cohort must be deemed treatable with an 8Fr IVUS from an anatomy and clinical safety perspective.

Intravascular ultrasound 0.035 PV catheter system

The investigational 0.035 PV IVUS catheter (Volcano Therapeutics, Rancho Cordova, CA) is an over the wire catheter-based ultrasound with an 8.2-French profile at the transducer end and 7.0-French shaft diameter. This is run through a 9-French place under surface ultrasound guidance in the common femoral artery. The working length of this catheter is 90 cm, with the ability to imaging a diameter up to 60 mm.7

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with an AAD or acute on chronic aortic dissection, with a new diagnosis of malperfusion syndrome (Malperfusion Primary Cohort), by meeting both of the following criteria:

  * Imaging findings indicating reduced flow to the Celiac Trunk, Superior mesenteric artery, either renal artery or either iliac artery
  * Clinical stigmata of end organ ischemia (abdominal pain, distended abdomen, oliguria/anuria, reduced pulses, signs of limb ischemia) correlating with imaging findings
* OR

  o Laboratory findings suggestive of end organ ischemia (lactic acidosis, elevated LFTs, Elevated Creatinine, Rhabdomyolysis, Electrolyte abnormalities) correlating with imaging findings
* Patients diagnosed with an AAD undergoing surgical repair without evidence of malperfusion syndrome preoperatively, but who develop malperfusion syndrome due to dynamic flow changes after true lumen flow is reinstituted intraoperatively as indicated by new clinical signs or new laboratory results meeting the following criteria (Malperfusion Secondary Cohort):

  * New Clinical signs include: Loss of femoral pulses, distended abdomen, reduced urine output, dusky/cold extremities
  * New Laboratory results include: Rising lactate (>50% above baseline), Rising Creatinine, Metabolic Acidosis, Rising LFTs
* Patients diagnosed with an AAD undergoing surgical repair without evidence of malperfusion syndrome preoperatively and postoperatively (No Malperfusion Cohort).

Exclusion Criteria:

* Subject has not been diagnosed with AAD, or acute on chronic aortic dissection
* Subject is not hemodynamically stable to undergo IVUS evaluation
* Subject has anatomy or pre-existing condition precluding safe use of IVUS evaluation
* Subject has a pre-existing condition that may explain evidence of malperfusion (i.e. Dialysis patient with severe renal stenosis).
* Subject or substitute decision maker has language barrier and no translator available at the time of obtaining informed consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 30 days
  Composite of all-cause in hospital mortality, acute kidney injury requiring new dialysis, mesenteric ischemia requiring intervention and major vascular complications.
Primary Effectiveness Endpoint | 30 days
  Composite of all-cause in hospital mortality, acute kidney injury requiring dialysis, mesenteric ischemia requiring surgical resection and major vascular complications.

SECONDARY OUTCOMES:
Secondary Effectiveness Endpoint | 30 days
  Composite of length of ICU stay and length of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Valdis, MD, FRCSC, Study Director — London Health Sciences Center , London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsai T, Nienaber CA, Isselbacher EM, Trimarchi S, Bossone E, Evangelista A, Oh JK, O'Gara P, Suzuki T, Hutchison S, Cooper JV, Meinhardt G, Myrmel T, Eagle KA, Froehlich J. Acute type A aortic dissection: does a primary tear in the aortic arch affect management and outcomes? Insights from the International Registry of Acute Aortic Dissection (IRAD). Circulation 2006; 114:432.8.
- [Result] HIRST AE Jr, JOHNS VJ Jr, KIME SW Jr. Dissecting aneurysm of the aorta: a review of 505 cases. Medicine (Baltimore). 1958 Sep;37(3):217-79. doi: 10.1097/00005792-195809000-00003. No abstract available. PMID 13577293
- [Result] Collins JS, Evangelista A, Nienaber CA, Bossone E, Fang J, Cooper JV, Smith DE, O'Gara PT, Myrmel T, Gilon D, Isselbacher EM, Penn M, Pape LA, Eagle KA, Mehta RH; International Registry of Acute Aortic Dissection (IRAD). Differences in clinical presentation, management, and outcomes of acute type a aortic dissection in patients with and without previous cardiac surgery. Circulation. 2004 Sep 14;110(11 Suppl 1):II237-42. doi: 10.1161/01.CIR.0000138219.67028.2a. PMID 15364869
- [Result] Yang B, Rosati CM, Norton EL, Kim KM, Khaja MS, Dasika N, Wu X, Hornsby WE, Patel HJ, Deeb GM, Williams DM. Endovascular Fenestration/Stenting First Followed by Delayed Open Aortic Repair for Acute Type A Aortic Dissection With Malperfusion Syndrome. Circulation. 2018 Nov 6;138(19):2091-2103. doi: 10.1161/CIRCULATIONAHA.118.036328. PMID 30474418
- [Result] Valdis M, Adams C, Chu MWA, Kiaii B, Guo L. Comparison of outcomes of root replacement procedures and supracoronary techniques for surgical repair of acute aortic dissection. Can J Surg. 2017 Jun;60(3):198-204. doi: 10.1503/cjs.009116. PMID 28570214
- [Result] Hagan PG, Nienaber CA, Isselbacher EM, Bruckman D, Karavite DJ, Russman PL, Evangelista A, Fattori R, Suzuki T, Oh JK, Moore AG, Malouf JF, Pape LA, Gaca C, Sechtem U, Lenferink S, Deutsch HJ, Diedrichs H, Marcos y Robles J, Llovet A, Gilon D, Das SK, Armstrong WF, Deeb GM, Eagle KA. The International Registry of Acute Aortic Dissection (IRAD): new insights into an old disease. JAMA. 2000 Feb 16;283(7):897-903. doi: 10.1001/jama.283.7.897. PMID 10685714
- [Result] Kpodonu J, Ramaiah VG, Diethrich EB. Intravascular ultrasound imaging as applied to the aorta: a new tool for the cardiovascular surgeon. Ann Thorac Surg. 2008 Oct;86(4):1391-8. doi: 10.1016/j.athoracsur.2008.06.057. PMID 18805213